CLINICAL TRIAL: NCT03112785
Title: Randomized Comparison Between the Fitmore and the CLS Stem in Patients Operated in One-stage Due to Bilateral Symptomatous Hip Disease
Brief Title: Fitmore Versus CLS Stem in Total Hip Arthroplasty. Bilateral One-stage Operations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Johan Karrholm, MD Professor in Orhopaedics, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fitmore2011
Record Dates: First submitted 2017-03-07; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Primary Hip Osteoarthritis; Secondary Hip Osteoarthritis Due to Idiopathic Femoral Head Necrosis, Childhood or Inflammatory Disease; Bilateral Hip Disease; Surgical Treatment
Keywords: Hip; Arthroplasty; Stem; Outcome
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: Patients with bilateral degenerative hip osteoarthritis are operated with a short stem total hip arthroplasty on one side and a conventional stem on the opposite side. Implant selection is randomised on the most symptomatic side, the second side receives the type of stem not used on the first one.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Total hip arthroplasty (Fitmore or CLS uncemented femoral stem made by Zimmer-Biomet, Warshaw, USA) — The most symptomatic side is randomised to one of the two stem types studied. If the patient has equal amount of symptoms on both sides, the one with most pronounced degenerative Changes on plain radiographs will be randomised. On the second side the type of stem not used on the first one will be inserted. All patients and allhip will receive the same type and design of cup.

SUMMARY:
Main question: Will use of a stem design that allows anatomical reconstruction of the hip joint improve the outcome in terms of hip function and patient satisfaction without causing any adverse effects?

Background: Total hip arthroplasty with use of the most well documented implants is a safe and cost-effective procedure. In the Swedish Hip Arthroplasty register the CLS stem has a 16 years implant survival of 97, 5 %. It is a classic design which requires resection of most of the neck. The stem also intrudes into the greater trochanter which in patients with certain types of proximal hip anatomy makes proper introduction of the stem difficult. Finally it has a standard stem length which will jeopardise future stem removal should there occur any late infection or instability problems.

Short uncemented stems have been introduced to enable a more anatomic reconstruction of the hip joint and to cause less invasion of the femoral canal to facilitate future revision should it be necessary. A more conservative resection of neck could also be of value to improve the clinical outcome by improved hip function and patient satisfaction.

Purpose of the present study and design: In a prospective study the clinical outcome, stem fixation and bone remodelling around a short stem (Fitmore) will be studied. The main focus will be to evaluate patient reported outcomes especially concerning function, over all satisfaction, pain and activity. All patients will receive the same cup (Trilogy). This cup is chosen because it has a very thorough documentation in prospective RSA studies and in the Swedish hip arthroplasty register. All cups will be supplied with insert made of high molecular polyethylene (Longevity).

Number of hips in the study: 44 consecutive cases

DETAILED DESCRIPTION:
Main question: Will use of a stem design that allows anatomical reconstruction of the hip joint improve the outcome in terms of hip function and patient satisfaction without causing any adverse effects?

Background: Total hip arthroplasty with use of the most well documented implants is a safe and cost-effective procedure. In the Swedish Hip Arthroplasty register the CLS stem has a 16 years implant survival of 97, 5 %. It is a classic design which requires resection of most of the neck. The stem also intrudes into the greater trochanter which in patients with certain types of proximal hip anatomy makes proper introduction of the stem difficult. Finally it has a standard stem length which will jeopardise future stem removal should there occur any late infection or instability problems.

Short uncemented stems have been introduced to enable a more anatomic reconstruction of the hip joint and to cause less invasion of the femoral canal to facilitate future revision should it be necessary. A more conservative resection of neck could also be of value to improve the clinical outcome by improved hip function and patient satisfaction.

Purpose of the present study and design: In a prospective study the clinical outcome, stem fixation and bone remodelling around a short stem (Fitmore) will be studied. The main focus will be to evaluate patient reported outcomes especially concerning function, over all satisfaction, pain and activity. All patients will receive the same cup (Trilogy). This cup is chosen because it has a very thorough documentation in prospective RSA studies and in the Swedish hip arthroplasty register. All cups will be supplied with insert made of high molecular polyethylene (Longevity).

Number of hips in the study: 44 consecutive cases

Methods: EQ-5D including VAS-scale to evaluate pain and over all satisfaction, (specific questionnaire concerning side preference), Harris Hip Score, DXA, radiostereometry and gait analysis.

A. Clinical parameters: EQ-5D form (including VAS for pain and satisfaction) is filled in by the patients. Harris Hip Score is filled in by the examiner. SF-36 and activity scale (UCLA) is filled in by the patient. Patients also fill in a study specific form including questions about hip preferred and a pain drawing. Clinical parameters will be studied preoperative after 1, 2, 5, 7 and 10 years.

B. Conventional radiography: Examinations will be done preoperatively, postoperatively, after 1, 2, 5, 7 and 10 years.

C. Computed tomography: Preoperatively, after 1 and 7 years.

D. DXA measurements: Postoperatively, after 6 months, 1, 2, 5, 7 and 10 years.

E. Radiostereometry: Postoperatively, after 3 and 6 months, 1, 2, 5, 7 and 10 years.

F. Gait analysis: 1 and 2 years.

Focus of interest:

A. Patient reported outcomes and especially Oxford Hip Score will constitute our primary outcome parameter.

B. Conventional radiography (preop with metallic indicator to determine magnification) will include AP, True lateral and pelvic view.

C. Computed Tomography will be done for preoperative planning in 3D (a new software has been developed). Preoperative planning in 3D will be done for booth types of prostheses. A prerequisite is that we have 3D-models available for all implants used in the study. Preoperative planning will also be done in 2D.

The CT-examinations will be also used to measure the anteversion of the femur (preoperatively) and of the femoral component (1 year exam). The influence of this parameter on clinical results and fixation will be studied. CT at 7 years will be compared with previous examinations to study development of any osteolysis.

D. DXA - studies will be done to study bone remodelling in terms of changes of bone mineral density around the implant. Both the femoral- and the acetabular side will be studied.

E. Radiostereometry. The cup will be marked during surgery. Model based RSA for the cup Component will also be used. On the femoral side the femoral head centre will be used to measure stem migration. Tantalum markers will be inserted into the acetabular bone and proximal femur.

Femoral component migration will be measured as translations of the femoral head centre in three directions (medial/lateral, proximal/distal, anterior/posterior). Implant migration between the 6 months and 1 year follow up will constitute our second outcome parameter.

Comments: From previous studies of uncemented stems it has been found that these implants often subside up to 1-2 mm and some even more during 6 months (rarely up to 1 year) and may thereafter become stable and at least according to conventional radiography achieve osseous fixation.

Two years after the operation patients will also be studied using dynamic RSA during active abduction and flexion. The aim is to study any-lift off during these motions. A new radiostereometric laboratory has been installed in 2010 which has facilitated these types of examinations.

In addition the fixation of the cup and wear (femoral head penetration) will be measured.

F. Gait analysis will be performed one and two years after the operation. The patients will be studied walking and when rising from a chair. This analysis will focus on flexion/extension, motions of the hip and the knee and the ground reacting forces. The ab/adduction movements over the hip during walking will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Hip anatomy suitable for the Fitmore stem according to preoperative planning
2. Males and females aged 35 to 75 years (with bilateral hip disease).
3. Primary osteoarthritis.
4. Secondary osteoarthritis due to idiopathic femoral head necrosis, childhood or inflammatory disease. -

Exclusion Criteria:

1. Treatment with Cortisol or known osteoporosis.
2. Low expected activity rate due to other diseases including any generalized joint disease.
3. Anatomy unsuitable for the Fitmore stem.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Preferred hip (the hip arthroplasty preferred by the patient, right or left side) | 2 years
  Study specific protocol in which the patient from a general view tics one of 3 options: left side, right side or no difference). In the term preferred view the patient is asked to consider all aspects they Think are important such as freedom from pain, mobility, function or any other type of discomfort.

SECONDARY OUTCOMES:
Stem subsidence (distal migration of the stem) | 2 years
  Stem subsidence in mm (distal migration of the femoral head center) measured with radiostereometry
Extent of radiolucent lines around the stem | 2 years
  Development of radiolucent lines in percent of total stem circumference as measured on conventional radiographs
Any new surgical procedure where the stem is removed or Exchanges (revision of the stem) | 2, 5 and 10 years
  Stem Exchange or removal due to loosening, dislocation or periprostheic fracture

CONTACTS AND LOCATIONS:
Overall Officials: Johan N Kärrholm, MD, Professor, Principal Investigator — Sahlgrenska University Hospital

IPD SHARING:
Plan to Share IPD: No